CLINICAL TRIAL: NCT01792193
Title: Quantitative Analysis of Gut-derived Neuropeptides in Cerebrospinal Fluid (CSF) of Patients With Parkinson's Disease and Healthy Controls
Brief Title: Gut-derived Neuropeptides in Cerebrospinal Fluid of Patients With Parkinson's Disease and Healthy Controls
Status: Completed | Type: Observational
Sponsor: Dr. Marcus Unger (Other)
Responsible Party: Sponsor-Investigator, Dr. Marcus Unger, Consultant / Oberarzt der Klinik für Neurologie, Universität des Saarlandes
Organization: Universität des Saarlandes (Other)
Other Study IDs: Studie 139/12
Record Dates: First submitted 2013-02-08; First posted 2013-02-15 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — CSF and serum samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Parkinson's disease: Patients with Parkinson's disease
- Control: Healthy controls

SUMMARY:
In previous work, the investigators analyzed the concentration of gut-derived peptides (ghrelin, pancreatic polypeptide [PP]) in serum of patients with Parkinson's disease (PD). The investigators have shown that the secretion pattern differs between PD patients and controls. Beside ghrelin and pancreatic polypeptide other gut-derived peptides (e.g. Glucagon-like-Peptide 1[GLP-1], Amylin, etc.) might be relevant for PD as well. The rational to investigate gut-derived peptides in the neurological disorder Parkinson's disease (PD) is based on the following considerations:

* Receptors for gut-derived peptides are expressed in Central Nervous System (CNS) structures that are affected by the neurodegenerative process underlying Parkinson's disease
* Gut-derived peptides are involved in the modulation of higher brain functions (mood, cognition, reward-related behaviour) that are frequently altered in Parkinson's disease.
* The secretion of gut peptides is (co-)regulated by the vagal nerve that is dysfunctional in Parkinson's disease.
* Certain gut-derived peptides (ghrelin, GLP-1) stimulate neurogenesis and might be able to prevent cell death in neurodegenerative disorders, including Parkinson's disease.

Objective:

Collection of CSF and serum samples in a standardized way in order to quantitatively measure the concentration of gut-derived peptides (ghrelin, leptin, glucose-dependent insulinotropic peptide [GIP], GLP-1, amylin, PP, peptide YY [PYY], and insulin). Scientific questions:

1. Do CSF (and serum) concentrations of these gut peptides differ between PD patients and controls?
2. Do CSF (and serum) concentrations of the investigated peptides correlate with clinical and / or epidemiological characteristics of the investigated subjects (age, gender, BMI, disease duration, severity of motor impairments, presence of non-motor symptoms, co-morbidities, medication, etc.)?

ELIGIBILITY:
Main Inclusion Criteria:

* Informed consent to participate
* Capability to understand risks of study-related procedures
* For PD cohort: diagnosis of (idiopathic) Parkinson's disease

Main Exclusion Criteria:

* Pregnancy
* Subjects incompetent to provide informed consent
* Subjects that cannot undergo a lumbar puncture for medical reasons (thrombocytopenia, anticoagulation, increased cranial pressure)
* For control cohort: presence of a neurodegenerative disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
CSF and serum concentration of ghrelin, leptin, GIP, GLP-1, amylin, PP, PYY, and insulin | The outcome measure will be assessed only once, after an overnight fast between 7 and 8 AM. Study-related procedure will be performed on one singel day. There will be no follow-up.
  CSF and corresponding serum samples will be collected in the fasting state in the morning. A standardized collection of the samples is crucial to avoid potential confounders (daytime, metabolic state, etc.). Samples will be frozen immediately and kept at minus 20°C until analysis. Samples will be analysed using a multiplex approach.

CONTACTS AND LOCATIONS:
Locations (1):
- Saarland University, Homburg / Saar, Saarland, Germany